CLINICAL TRIAL: NCT02379663
Title: Efficacy and Safety for Prophylaxis of Deep Vein Thrombosis Following Total Hip Arthroplasty
Brief Title: Prophylaxis of Deep Vein Thrombosis Following Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-11-012
Record Dates: First submitted 2015-02-13; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthritis, Hip; Femur Head Necrosis; Femoral Neck Fractures
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis; Femoral Neck Fractures | interventions — Rivaroxaban; Enoxaparin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral direct Factor Xa inhibitor (Active Comparator): Rivaroxaban
  Interventions: Drug: Rivaroxaban
- Low molecular weight heparin (Active Comparator): Enoxaparin
  Interventions: Drug: Enoxaparin
- Normal Saline (Placebo Comparator): Normal Saline
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban was taken orally in a dosage of 10mg once daily
  Arms: Oral direct Factor Xa inhibitor
Drug: Enoxaparin — Enoxaparin was injected subcutaneously in a dosage of 40mg once daily
  Arms: Low molecular weight heparin
Other: Normal saline — subcutaneous injection of 1 cc of normal saline once daily
  Arms: Normal Saline

SUMMARY:
This prospective study compares an oral direct factor Xa inhibitor with LMWH for thromboprophylaxis in the patients undergoing THA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female without childbearing potential aged ≥20 years who were scheduled for elective primary THA

Exclusion Criteria:

* recent history of active bleeding or VTE
* known genetic disorder associated with bleeding tendency or any condition related with an increased risk of bleeding
* persistent blood pressure of ≥160mmHg systolic and/or ≥100 mmHg diastolic at baseline
* myocardial infarction or cerebrovascular accident within three months of the scheduled surgery
* major surgery in the prior three months
* renal insufficiency with a creatinine clearance <60mL/min , hepatic failure combined with coagulopathy, or thrombocytopenia (platelets < 100,000/mm³), or planned indwelling epidural catheter for > 6 hours after the end of surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Major wound complication | 2 weeks
  hematoma : size, site woozing : frequency, amount, dressing change count infection : culture